CLINICAL TRIAL: NCT05967078
Title: ExerG: Video Game-based Physical Cognitive Training for Patients: a Usability Study
Acronym: ExerGetic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frank Behrendt (Other)
Collaborators: Innosuisse - Swiss Innovation Agency (Other)
Responsible Party: Sponsor-Investigator, Frank Behrendt, Sponsor-Investigator, Reha Rheinfelden
Organization: Reha Rheinfelden (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-00559
Record Dates: First submitted 2023-06-19; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Gait Disorders, Neurologic; Gait Disorders in Old Age; Gait Disorder, Sensorimotor; Balance; Distorted; Functional Movement Disorder; Visual Disorder; Cognitive Impairment
MeSH Terms: conditions — Gait Disorders, Neurologic; Conversion Disorder; Vision Disorders; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): The device under investigation is the ExerCube training software licence provided by Sphery (https://sphery.ch/exercube/). The ExerCube training software licence is an exergame training product that includes immersive mixed-reality training programs (or video games) for patients. Depending on the patient's training requirements, the therapists can choose from the training program repertoire. The ExerCube supporting material for safety consisting of a harness and an over-head gantry system ensures a safe training environment and prevents patients from falling.
  Interventions: Device: ExerG

INTERVENTIONS:
Device: ExerG — The intervention for primary end users (PEU, (patients)) includes the performance of two training rounds with the device. The first round includes a predefined training sequence, whereas the second round is a training sequence defined by the therapist.
  For the secondary end user group (SEU, (therapists)), there are two study visits. At their first visit they get an introduction and training on how to use the system. At their second visit, SEU will have to prepare the device (switch on hard- and software) and guide the patient through the training.
  Other Names: ExerG training software licence

SUMMARY:
Video game-based training programs, in the following referred to as "exergames" are an innovative digital training approach to simultaneously train physical and cognitive functions and increase training motivation for various populations. Patients who are differently limited in their physical and cognitive performance due to a decline in functioning can profit from a motivating and combined physical-cognitive training approach. An interdisciplinary team of movement scientists, sports and training experts, as well as game and industrial designers developed an innovative and immersive video game-based training product for patients - the ExerCube training software licence. The exergame development focused on a user-centred process together with the target population.

The ExerCube training software licence is an exergame training product that includes immersive mixed-reality training programs (or video games) for patients. Depending on the patient's training requirements, the therapists can choose from the training program repertoire. The patients control the training program (or video game) by specific (whole) body movements. To present the virtual training programs from the ExerCube training software licence in the physical environment, the ExerCube hardware and harness system is used to serve as a physical training room. It allows the virtual video game environment to be presented in the physical world.

This summative usability study aims to assess the training system's safety, usability and validate the user experience.

Primary end-users (defined as patients aged 18 and above) and secondary end-users (defined as sports scientists, training therapists or physiotherapists/occupational therapists with a focus on sports/training therapy) will test and review the system in different testing scenarios.

ELIGIBILITY:
Inclusion Criteria:

Primary end users:

* in-/ or outpatients of the Reha Rheinfelden
* Ability to speak and comprehend German and to understand the digitally transmitted training instructions
* Body height ≥ 160 cm or ≤ 200 cm according to hardware specifications
* Body weight ≤ 120 kg
* Able to execute the movements of the video game-based training (being able to transfer from a sitting to a standing position and maintain the standing position without assistance for ≥ 2 minutes)

Secondary end users:

* therapists (physiotherapist, occupational therapist, sport scientist, sport therapist, psychologists) working in the area of rehabilitation and prevention
* ≥ 21 years of age
* Bachelor's degree (scientists) or completed education as therapist

Exclusion Criteria:

Primary end users

* Cognitive impairment as defined by a Mini Mental State Examination (MMSE) score of ≤ 18
* Severe visual, neurological, cardiorespiratory, psychiatric, or orthopedic impairments which reduce the person's capability of following the instructions or to play the game
* Recently occurred epileptic seizures (in the past 3 months)
* Recent surgery/fractures/surgical interventions/joint replacement and malignancy (in the past 3 months)
* Physical conditions in which a correct wearing of the Safety harness is not possible or could cause pain or health problems (e.g. skin lesions, open wounds, known pregnancy, severe osteoporosis)
* Joint contractures (e.g. shoulder, knee, hip) that could lead to limitations during end-user evaluation of the ExerCube.
* Severe neurologic illness (e.g., strong epilepsy, advanced parkinson's syndrome, condition after severe stroke)
* Severe psychiatric illness (e.g., pronounced paranoid states, severe depression)
* Terminal illness (prognosis < 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Usability: performance rate | 1 day
  The acceptance of the device is rated based on the observation protocol that is completed by the study moderator during the training session. Each participant will have a list of tasks to be completed per session/ training round.
  Primary end users (PEU): acceptance criteria for performance = correct task performance "yes" ≥ 85%, skipped tasks < 20%
  Secondary end users (SEU): acceptance criteria for performance = task performed correctly or with hesitant behaviour ≥ 85%, task not performed or with difficulties and failures < 15%
Usability: Number of participants with no need for support | 1 day
  The acceptance of the device is rated based on the observation protocol that is completed by the study moderator during the training session. Each participant will have a list of tasks to be completed per session/ training round.
  Primary end users (PEU): acceptance criteria for comprehensibility = very good or good comprehension about how to perform the task ≥ 85%
  Secondary end users (SEU): acceptance criteria for support = task performed without support ≥ 85%, support needed to be able to complete the task < 15%
Usability: exercise execution | 1 day
  The acceptance of the device is rated based on the observation protocol that is completed by the study moderator during the training session. Each participant will have a list of tasks to be completed per session/ training round.
  Primary end users (PEU):
  - acceptance criteria for exercise execution = very good or good exercise/ movement execution ≥ 85%
Usability: Number of (serious) adverse events | 1 day
  (Serious) Adverse Events: acceptance criteria of occurrence of related adverse events should not exceed 10%.
Usability: device deficiencies | 1 day
  Acceptance criteria for occurence of any device deficiencies encountered during study visits is set to <10%.

SECONDARY OUTCOMES:
Usability: Player Experience | 1 day
  Primary end users (PEUs): The user experience will be assessed with the Player Experience Inventory (PXI), a 30 item questionnaire containing 10 different constructs to measure different aspects of player experience (three items per construct). All items are rated on a 7-point Likert scale (scale range: -3 to 3 points, maximal score = +90; minimal score: -90).
Usability: System Usability | 1 day
  Secondary end users (SEUs): The System Usability Scale (SUS) will be completed by secondary end users to evaluate the perceived usability. SUS assesses perceived effectiveness (can users successfully achieve their objectives), information quality (how much effort and resource is expended in achieving those objectives) and general satisfaction (was the experience satisfactory). The SUS hast 10 items that can be rated on a 5-point likert scale. The items will be scored as follows:
  1. For odd-numbered items, user response-1. For even-numbered items 5-user response. This scales all values from 0 to 4 (with four being the most positive response). Ref: Jeff Sauro, measuring usability
  2. Add up the converted responses for each user and multiply that total by 2.5 (to convert the range of possible values from 0 to 100 instead of from 0 to 40)
Perceived physical and mental exertion/ effort | 1 day
  Perceived physical exertion during the training will be assessed with the Borg-category rating 10 (Borg CR10; scale range from 0= no exertion at all, 10= maximal level of exertion).
  Perceived mental effort will be assessed from primary end users with the Paas mental effort scale (Paas, 1992) ranging from 1= very, very low mental effort, 9=very, very high mental effort.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Behrendt, PhD, Principal Investigator — Reha Rheinfelden
Locations (1):
- Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No